CLINICAL TRIAL: NCT07227675
Title: Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional MR Continued Access Study
Brief Title: Cardiovascular Outcomes Assessment of the MitraClip Percutaneous Therapy for Heart Failure Patients With Functional MR
Acronym: COAPT CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11- 512
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Mitral Regurgitation; Mitral Valve Regurgitation
Keywords: Functional Mitral Regurgitation; Mitral Valve Regurgitation; Symptomatic Heart Failure; COAPT CAS
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- The MitraClip NT Device (Experimental): The MitraClip NT System comprises the MitraClip NT Clip Delivery System
  Interventions: Device: MitraClip® NT System

INTERVENTIONS:
Device: MitraClip® NT System — The MitraClip NT System is intended to treat heart failure patients with symptomatic ischemic or non-ischemic functional MR

SUMMARY:
The COAPT Continued Access Study (CAS) is an extension of the COAPT RCT under the same IDE (G120024). COAPT CAS was a single-arm, prospective, multicenter continued access registry that enrolled heart failure patients with secondary mitral regurgitation who remained symptomatic despite optimal guideline-directed medical therapy (GDMT). The objective of the COAPT CAS is to continue the evaluation of safety and effectiveness of the MitraClip NT System under more "real world" conditions in patients who meet the COAPT inclusion/exclusion criteria and who have national Medicare coverage by the Centers for Medicare and Medicaid Services (CMS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have national Medicare coverage by CMS
* Symptomatic functional MR (≥3+) due to cardiomyopathy of either ischemic or non-ischemic etiology
* Subject has been adequately treated per applicable standards, including for coronary artery disease, left ventricular dysfunction, mitral regurgitation and heart failure
* Subject has had at least one hospitalization for heart failure in the 12 months prior to subject registration and/or a corrected BNP ≥300 pg/ml or corrected NT-proBNP ≥1500 pg/ml
* New York Heart Association (NYHA) Functional Class II, III or ambulatory IV
* Surgery will not be offered as a treatment option and medical therapy is the intended therapy for the subject
* Left Ventricular Ejection Fraction (LVEF) is ≥20% and ≤50%
* Left Ventricular End Systolic Dimension (LVESD) is ≤70 mm

Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization
* Coronary artery bypass grafting (CABG) within prior 30 days
* Percutaneous coronary intervention within prior 30 days
* Tricuspid valve disease requiring surgery
* Aortic valve disease requiring surgery
* Chronic Obstructive Pulmonary Disease (COPD) requiring continuous home oxygen therapy or chronic outpatient oral steroid use
* Cerebrovascular accident within prior 30 days
* Severe symptomatic carotid stenosis (> 70% by ultrasound)
* Carotid surgery within prior 30 days
* Mitral valve orifice area < 4.0 cm2
* Leaflet anatomy which may preclude MitraClip implantation, proper MitraClip positioning on the leaflets or sufficient reduction in MR by the MitraClip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Safety end point: Freedom from death | through 5 years
Safety end point: Freedom from Myocardial Infarction (MI) | through 5 years
Safety end point: Freedom from stroke | through 5 years
Safety end point: Heart Failure Hospitalization | through 5 years
Recurrent Heart Failure Hospitalization | through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mack, MD, Principal Investigator — Baylor Health Care System; William T Abraham, MD, Principal Investigator — The Ohio State University Heart Center; JoAnn Lindenfeld, MD, Principal Investigator — Vanderbilt University Medical Center; Gregg W Stone,, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (32):
- United States (32):
  - Scripps Green Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Mount Sinai Medical Center, Miami, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Hospital Atlanta, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - Seton Medical Center Austin, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - The heart hospital baylor plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia